CLINICAL TRIAL: NCT04929743
Title: Randomized Clinical Trial to Evaluate the Predictability and Evolution of Extra-short 5.5 mm Dental Implants Splinted in Partial or Complete Prostheses
Brief Title: Randomized Clinical Trial to Evaluate the Predictability of 5.5 mm Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTI_02_EC/20/4.5
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 5.5 mm implants (Experimental)
  Interventions: Device: BTI Implant
- >6.5 mm implants (Active Comparator)
  Interventions: Device: BTI Implant

INTERVENTIONS:
Device: BTI Implant — Placement of dental implants of 5.5 vs >6.5 mm length

SUMMARY:
The main aim of this clinical trial is to analyze the survival rate of short-length implants (<4.5 mm) in partial edentulism subjects. 6.5 mm length implants will be used as control arm. Additionally, others clinical parameters (marginal bone loss and prosthetic associated complications) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical indication to place a prosthetic bridge supported by a maximum of 4 implants in the posterior sectors
* Bone height in the area of interest sufficient to place implants 6.5mm length dental implants
* Availability to be observed during the follow-up period
* Signature of the informed consent

Exclusion Criteria:

* Need to perform bone augmentation surgery prior to implant placement surgery
* Smokers (> 10 cigarettes per day)
* Patients with poorly controlled diabetes
* Patients on chronic treatment with non-steroidal anti-inflammatory drugs
* Patients receiving oral or intravenous bisphosphonates
* Patients under chemotherapy or radiotherapy treatment
* Patients receiving systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Survival of implants | 1 year
  Survival of implants at one year post-implantation

SECONDARY OUTCOMES:
Marginal bone loss | 1 year
  Marginal bone loss at one year post-implantation
Incidence of bleeding on probing | 1 year
Incidence of prosthetic or implant complications | 1 year
Probing pocket depth | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Eduardo Anitua, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided